CLINICAL TRIAL: NCT03943459
Title: Serum Concentration and Gene Expression of Sirtuin-1 and Advanced Glycation End-products in Postmenopausal Women With Atherosclerotic Coronary Disease After Administration of Atorvastatin and Supplementation With Quercetin: Randomized Trial
Brief Title: Sirtuin-1 and Advanced Glycation End-products in Postmenopausal Women With Coronary Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, ANTONIO DE PADUA MANSUR, Associate Professor, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 408720/2018-2
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease Progression
Keywords: coronary artery disease; sirtuins; Receptor for Advanced Glycation End Products; women; quercetin; atorvastatin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Quercetin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): 20 Patients on placebo
- Atorvastatin (No Intervention): 20 patients treated with atorvastatin 80 mg/day
- Quercetin (Experimental): 20 patients treated with quercetin 500 mg/day
  Interventions: Drug: Quercetin

INTERVENTIONS:
Drug: Quercetin — Quercetin 250 mg BID
  Other Names: Atorvastatin
  Arms: Quercetin

SUMMARY:
Higher consumption of fruits and vegetables promote greater availability of phenolic compounds and these compounds were associated with vascular health. Quercetin, a phenolic compound, is the most abundant natural antioxidant belonging to the group of flavonoids. Quercetin improved lipoprotein metabolism, had antioxidant capacity, produced vasodilating substances in the vascular endothelium and reduced platelet aggregability. Likewise, statins are medications known to reduce cardiovascular events in women with coronary disease by reducing serum LDL-cholesterol. Therefore, a number of metabolic pathways are responsible for vascular health. The serum concentration and gene expression of sirtuin 1 (Sirt1) and RAGE soluble (sRAGE) are directly associated with vascular protection. This study will analyse the influence of atorvastatin and quercetin on serum concentrations and gene expression of Sirt1 and sRAGE in postmenopausal women with stable coronary artery disease.

DETAILED DESCRIPTION:
Higher consumption of fruits and vegetables promote greater availability of phenolic compounds and these compounds were associated with vascular health. Quercetin, a phenolic compound, is the most abundant natural antioxidant belonging to the group of flavonoids. Quercetin improved lipoprotein metabolism, had antioxidant capacity, produced vasodilating substances in the vascular endothelium and reduced platelet aggregability. Likewise, statins are medications known to reduce cardiovascular events in women with coronary artery disease (CAD) by reducing serum LDL-cholesterol. Therefore, a number of metabolic pathways are responsible for vascular health. The serum concentration and gene expression of sirtuin 1 (Sirt1) and RAGE soluble (sRAGE) are directly associated with vascular protection. This study will analyse the influence of atorvastatin and quercetin on serum concentrations and gene expression of Sirt1 and sRAGE in postmenopausal women with stable coronary artery disease and also the correlation between the changes in serum concentration of Sirt1 and sRAGE and the changes in lipid profile, inflammatory biomarkers and sex hormones in response to these drugs. This is a 60-day randomized, double blind, placebo-controlled study in 60 postmenopausal women with CAD, divided into three groups with 20 women each: Group 1 - Quercetin (500 mg / day); Group 2 - atorvastatin (80 mg / day): Group 3 - control.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women,
* angiographic documented coronary artery disease,
* stable coronary artery disease

Exclusion Criteria:

* BMI <18,1 Kg/m2,
* smoking,
* hypo or hyperthyroidism,
* rheumatic disease,
* use of alcohol,
* hepatic failure,
* renal failure
* hormone replacement therapy
* use of insulin

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Sirtuin-1 | 60 days
  serum concentration of sirtuin-1
Soluble receptor for advanced glycation end products | 60 days
  serum concentration of soluble receptor for advanced glycation end products

CONTACTS AND LOCATIONS:
Overall Officials: Antonio P Mansur, PhD, Principal Investigator — InCor Heart Institute
Locations (1):
- INCOR - Heart Institute, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.